CLINICAL TRIAL: NCT01101893
Title: A Phase I, Open Label, Single Sequence, Drug Interaction Study Evaluating Plasma GSK2248761 and Raltegravir Pharmacokinetics in Healthy Adult Subjects.
Brief Title: A Drug Interaction Study Evaluating GSK2248761 and Raltegravir Pharmacokinetics in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: E.D. Derilus; Clinical Disclosure Advisor, GSK Clinical Disclosure
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 113392
Record Dates: First submitted 2010-04-08; First posted 2010-04-12 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Infection, Human Immunodeficiency Virus
Keywords: GSK2248761, raltegravir, drug interaction, pharmacokinetics
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — Raltegravir Potassium; IDX 899

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Period 1 (Experimental): In period 1 all subjects will receive Raltegravir 400mg q12h from Day 1 to Day 5
  Interventions: Drug: Raltegravir
- Period 2 (Experimental): In period 2 all subjects will receive GSK2248761 200mg q24h from Day 1 to Day 5.
  Interventions: Drug: GSK2248761
- Period 3 (Experimental): Day 1 of Period 3 will be the day after Day 5 of Period 2. Subjects will receive GSK2248761 200mg q24h + raltegravir 400mg q12h from Day 1 to Day 5.
  Interventions: Drug: GSK2248761 + Raltegravir

INTERVENTIONS:
Drug: Raltegravir — raltegravir 400mg q12h x 5 days (Reference Treatment)
  Arms: Period 1
Drug: GSK2248761 — GSK2248761 200mg q24h x 5 days (Reference Treatment)
  Arms: Period 2
Drug: GSK2248761 + Raltegravir — GSK2248761 200mg q24h + raltegravir 400mg q12h x 5 days (Test Treatment)
  Arms: Period 3

SUMMARY:
In this study, approximately 16 subjects will receive raltegravir 400mg twice daily for 5 days (Treatment A) followed by a washout period. In Period 2, subjects will receive GSK2248761 200mg once daily for 5 days (Treatment B). There will be no wash out between Period 2 and 3. Subjects will then be administered raltegravir 400mg twice daily in combination with GSK2248761 200mg once daily (Treatment C) for 5 days. Subjects will be housed in the unit for the duration of the study. Safety evaluations and serial PK samples will be collected during each treatment period. A follow-up visit will occur 7-14 days after the last dose of study drug.

DETAILED DESCRIPTION:
ViiV Healthcare is the new sponsor of this study, and GlaxoSmithKline is in the process of updating systems to reflect the change in sponsorship.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, vital signs, laboratory tests, and ECGs. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Male or female between 18 and 50 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of non-childbearing potential (i.e., physiologically incapable of becoming pregnant) including any female who:
* Is pre-menopausal with a documented bilateral tubal ligation, bilateral oophorectomy (removal of the ovaries) or hysterectomy, or is post-menopausal defined as 12 months of spontaneous amenorrhea. A follicle stimulating hormone (FSH) level will be performed to confirm a post-menopausal status. For this study, FSH levels > 40 MlU/ml is confirmatory.
* Male subjects must agree to use one of the contraception methods listed in Section 8.1 of the study protocol. This criterion must be followed from the time of the first dose of study medication until the follow-up visit.
* Body weight greater than or equal to 50 kg for men and greater than or equal to 45 kg for women and body mass index (BMI) within the range 18.5-31.0 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* As a result of the medical interview, physical examination, or screening investigations, the Investigator considers the subject unfit for the study.
* The subject has a positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* Unwilling to refrain from the use of illicit drugs and adhere to other protocol-stated restrictions while participating in the study.
* History of regular alcohol consumption within 6 months of the study defined as: An average weekly intake of >14 drinks/week for men or >7 drinks/week for women. Note: One drink is equivalent to (12 g alcohol) = 5 ounces (150 ml) of wine or 12 ounces (360 ml) of beer or 1.5 ounces (45 ml) of 80 proof distilled spirits.
* Unwilling to abstain from alcohol for 48 hours prior to the start of dosing until collection of the final pharmacokinetic sample during each treatment period.
* History or regular use of tobacco- or nicotine-containing products within 3 months prior to screening.
* History/evidence of symptomatic arrhythmia, angina/ischemia, coronary artery bypass grafting (CABG) surgery or percutaneous transluminal coronary angioplasty (PCTA) or any clinically significant cardiac disease.
* History/evidence of clinically significant pulmonary disease.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Subjects with a pre-existing condition interfering with normal gastrointestinal anatomy or motility, hepatic and/or renal function, that could interfere with the absorption, metabolism, and/or excretion of the study drugs. Subjects with a history of cholecystectomy should be excluded.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation. In addition, if heparin is used during PK sampling, subjects with a history of sensitivity to heparin or heparin-induced thrombocytopenia should not be enrolled.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.

Note: this does not include plasma donation.

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A positive test for HIV antibody.
* AST, ALT, alkaline phosphatase and bilirubin greater than or equal to 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Pregnant females as determined by positive serum hCG test at screening or prior to dosing.
* Lactating females.
* The subject's systolic blood pressure is outside the range of 90-140mmHg, or diastolic blood pressure is outside the range of 45-90mmHg or heart rate is outside the range of 50-100bpm for female subjects or 45-100 bpm for male subjects at Screening and predose Day 1.

Cardiac conduction abnormalities denoted by any of the following on a single 12-lead ECG at screening or predose Day 1 (a single repeat is allowed for eligibility determination) Evidence of previous myocardial infarction (Does not include ST segment changes associated with repolarization).

Any conduction abnormality (including but not specific to left or right complete bundle branch block, AV block [2nd degree or higher], Wolf Parkinson White [WPW] syndrome).

Sinus Pauses > 3 seconds. Any significant arrhythmia which, in the opinion of the principal investigator and GSK medical monitor, will interfere with the safety for the individual subject.

Non-sustained or sustained ventricular tachycardia (greater than or equal to 3 consecutive ventricular ectopic beats)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2010-04; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Plasma raltegravir steady-state CL/F, AUC(0-tau), Cmax, tmax, Ctau, and Cmin following administration of raltegravir 400mg q12h for 5 days and following co-administration with GSK2248761 200mg q24h for 5 days. | 5 days
Plasma GSK2248761 steady state PK parameters, including CL/F, AUC(0-tau), Cmax, tmax, Ctau, & Cmin following administration of GSK2248761 200mg q24h for 5 days & following co-administration of raltegravir 400 mg q12h & GSK2248761 200 mg q24h for 5 days | 5 days

SECONDARY OUTCOMES:
Safety and tolerability parameters, including adverse event, concurrent medication, clinical laboratory, ECG, and vital signs assessments | approximately 34 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Buffalo, New York, United States

REFERENCES:
- [Derived] Piscitelli S, Kim J, Gould E, Lou Y, White S, de Serres M, Johnson M, Zhou XJ, Pietropaolo K, Mayers D. Drug interaction profile for GSK2248761, a next generation non-nucleoside reverse transcriptase inhibitor. Br J Clin Pharmacol. 2012 Aug;74(2):336-45. doi: 10.1111/j.1365-2125.2012.04194.x. PMID 22288567